CLINICAL TRIAL: NCT03109704
Title: The Immediate Effects of a Seated Versus Supine Upper Thoracic Spine Thrust Manipulation Compared to Sham Manipulation in Individuals With Subacromial Pain Syndrome: A Randomized Controlled Trial
Brief Title: Thoracic Spine Thrust Manipulation Compared to Sham Manipulation in Individuals With Subacromial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sacred Heart University (Other)
Collaborators: Nova Southeastern University (Other)
Responsible Party: Principal Investigator, Jason Grimes, PT, PhD, OCS, ATC, Clinical Assistant Professor, Sacred Heart University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 151119A
Record Dates: First submitted 2017-03-29; First posted 2017-04-12 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-03

CONDITIONS: Subacromial Impingement; Subacromial Impingement Syndrome
Keywords: scapular kinematics; thoracic spine; thrust manipulation
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Intervention Model Description: randomized controlled trial, 3 groups which includes a sham comparator
Who Masked: Participant
Masking Description: participants were made aware of the 3 different interventions being investigated but were not told which technique they were assigned to receive
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supine thrust manipulation (Experimental): The supine upper thoracic spine thrust manipulation will be performed two times, regardless of joint cavitation.
  Interventions: Procedure: Supine upper thoracic spine thrust manipulation
- Seated thrust manipulation (Experimental): The seated upper thoracic spine thrust manipulation will be performed two times, regardless of joint cavitation.
  Interventions: Procedure: Seated upper thoracic spine thrust manipulation
- Sham manipulation (Sham Comparator): The sham manipulation will be performed two times.
  Interventions: Procedure: Sham manipulation

INTERVENTIONS:
Procedure: Supine upper thoracic spine thrust manipulation — The supine thrust manipulation will target the upper thoracic spine and will be performed as previously described. The patient will be asked to lace his or her fingers behind the neck and bring his or her elbows close together in front of the chest. The therapist will place one hand just below the targeted upper thoracic region (at either the T3 or T4 level) using a pistol grip or loose fist to make contact with both transverse processes of the T3 or T4 vertebrae. The therapist will then use his or her body to push down through the patient's upper arms to provide a high-velocity, low-amplitude thrust in the anterior-to-posterior direction.
  Arms: Supine thrust manipulation
Procedure: Seated upper thoracic spine thrust manipulation — The seated thrust manipulation will target the cervicothoracic junction with the patient sitting with fingers laced behind the neck. The therapist will stand behind the patient and thread his or her arms through the patient's arms and clasp his or her hands near the C7-T1 level. The therapist will make contact with his or her chest against the patient's upper thoracic region to serve as a fulcrum. The patient will then be instructed to take a deep breath, and upon exhalation the therapist will apply a high-velocity, low-amplitude distraction thrust in a cephalad direction.
  Other Names: C-T junction distraction manipulation
  Arms: Seated thrust manipulation
Procedure: Sham manipulation — The sham manipulation will be performed with the patient and the examiner positioned in the same manner as for the seated manipulation, however the examiner will apply only minimal pressure to maintain physical contact and "skin lock" with the patient. The examiner will then move the patient through the same range of motion but deliver no manipulative thrust.
  Arms: Sham manipulation

SUMMARY:
This study evaluates the immediate and short-term effects of a supine upper thoracic spine thrust manipulation, seated upper thoracic spine thrust manipulation, and sham manipulation for individuals with subacromial pain syndrome. The participants were randomized to receive one of the three interventions and baseline measures for the dependent variables were repeated immediately after the delivery of the intervention.

DETAILED DESCRIPTION:
Thoracic spine thrust manipulation has been shown to be effective in reducing pain and improving function in individuals with subacromial pain syndrome (subacromial impingement). It remains unknown if individuals respond differently to different manipulation techniques. This study examines the immediate effects on pain and short-term effects on pain and function using the Penn Shoulder Score (PSS) as well as the immediate effects on scapular kinematics (upward rotation and posterior tilt, specifically), pectoralis minor muscle length, and scapulothoracic muscle force production for the middle trapezius, lower trapezius, and serratus anterior.

ELIGIBILITY:
Inclusion Criteria:

* currently experiencing shoulder pain for less than 6 months
* at least 3 of the following findings: 1) pain localized to the proximal anterolateral shoulder region, 2) positive Neer or Hawkins-Kennedy impingement test, 3) pain with active shoulder elevation (which may include a painful arc), 4) active shoulder abduction ROM of at least 90°, 5) passive shoulder external rotation ROM of at least 45°, and 6) pain with isometric resisted abduction or external rotation

Exclusion Criteria:

* signs of a complete rotator cuff tear
* significant loss of glenohumeral motion
* acute inflammation
* cervical spine-related symptoms including a primary complaint of neck pain, signs of central nervous system or cervical nerve root involvement, or reproduction of shoulder or arm pain with cervical rotation, axial compression, or Spurling test
* previous neck or shoulder surgery
* positive apprehension test or relocation test
* history of shoulder fracture or dislocation
* history of nerve injury affecting upper extremity function
* any contraindication for thrust manipulation to the thoracic spine including osteoporosis, fracture, malignancy, systemic arthritis, or infection
* fear or unwillingness to undergo thoracic spine manipulation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-10-24 (Actual); Study Completion 2016-10-26 (Actual)

PRIMARY OUTCOMES:
Change in Penn Shoulder Score (PSS) from baseline to 48 hours | baseline and 48 hours after intervention
  The Penn Shoulder Score is a 100-point shoulder-specific questionnaire with three subscales: self-reported pain, function, and satisfaction with current use of the shoulder. The scores from the subscales are summed to determine the total score with the pain subscale score ranging from 0-30, function subscale score ranging from 0-60, and satisfaction subscale score ranging from 0-10. The total maximum score of 100 points indicates high function, low pain, and high satisfaction with the shoulder.
Change in pain | baseline and 1 minute after intervention
  Pain will be measured using the verbal numeric rating scale (VNRS). Participants will be asked to rate their pain on a 0-10 scale with 0 indicating no pain and 10 indicating the worst pain imaginable. This pain rating will be obtained during active elevation of the arm in the scapular plane.

SECONDARY OUTCOMES:
Change in scapular upward rotation active range of motion (ROM) | baseline and 1 minute after intervention
  The participant will start with the involved arm at the side of the body. The investigator will confirm the location of the scapular plane by placing the subject's arm at an angle 40 degrees anterior from the frontal plane as measured with a standard goniometer. The digital inclinometer will be zeroed on a horizontal surface and then placed along the scapular spine of the involved arm. The initial reading from the inclinometer on the scapular spine with the arm at the side of the body will be recorded. The subject will then be instructed to elevate the arm in the scapular plane as high as he/she can go. The final reading from the inclinometer will then be recorded at the end of the subject's maximal arm elevation. The total amount of scapular upward rotation will be calculated as the change score by taking the difference between the final and initial readings. Downward rotation would be recorded as negative values and upward rotation would be recorded as positive values.
Change in scapular posterior tilt active ROM | baseline and 1 minute after intervention
  The participant will start with the test arm at the side of the body. The digital inclinometer will be zeroed on a vertical surface and then placed vertically along the posterior surface of the medial border of the scapula, using the root of the scapular spine and the inferior angle of the scapula as landmarks as previously described. The initial reading from the inclinometer with the arm at the side of the body will be recorded. The subject will then be instructed to elevate the arm in the scapular plane as high as he/she can go. The final reading from the inclinometer will then be recorded at the end of the subject's maximal arm elevation. The total amount of scapular posterior tilt will be calculated as the change score by taking the difference between the final and initial readings. Anterior tilt would be recorded as negative values and posterior tilt would be recorded as positive values.
Change in scapular upward rotation passive ROM | baseline and 1 minute after intervention
  Measurements will be made with the subject in standing. The participant will start with the involved arm at the side of the body. The digital inclinometer will be zeroed and positioned as described for the measure of upward rotation active ROM. The initial reading from the inclinometer will be recorded. The examiner can then passively elevate the humerus in the scapular plane to end-range elevation, producing passive upward rotation of the scapula. The examiner will move the subject's arm through the full available elevation ROM passively for two consecutive trials. At the point of maximal passive arm elevation on the second repetition, the inclinometer will again be placed along the scapular spine to obtain a measurement of upward rotation passive ROM. The total amount of scapular upward rotation passive ROM will be calculated as the change score by taking the difference between the final and initial readings.
Change in scapular posterior tilt passive ROM | baseline and 1 minute after intervention
  Measurements will be made with the subject standing. The digital inclinometer will be zeroed and positioned as described for the measure of posterior tilt active ROM. The initial reading from the inclinometer will be recorded with the subject's arm at the side of the body. The examiner can then passively elevate the humerus in the scapular plane to end-range elevation, producing passive posterior tilt of the scapula. The examiner will move the subject's arm through the full, available elevation ROM passively for two consecutive trials. At the point of maximal passive arm elevation on the second repetition, the inclinometer will again be placed along the posterior surface of the medial border of the scapula to obtain a measurement of posterior tilt passive ROM. The total amount of scapular posterior tilt passive ROM will be calculated as the change score by taking the difference between the final and initial readings.
Change in pectoralis minor muscle length | baseline and 1 minute after intervention
  Performed as described previously by Borstad. A tape measure will be used to measure the linear distance in cm between the anterior-inferior edge of the 4th rib one finger width lateral to the sternum and the medial-inferior aspect of the coracoid process of the scapula. This measurement will be completed while the subject is standing in their usual resting position.
Change in middle trapezius force production | baseline and 1 minute after intervention
  A handheld dynamometer (HHD) (Hoggan MicroFET2) will be used to assess force production in standard manual muscle test (MMT) position using a "make test" as previously described. The "make test" will require the examiner to instruct the subject to slowly push into the HHD and increase their force production to a maximal level over a 5-second period of time. Prior to maximal isometric testing, a sub-maximal (50%) effort trial will be performed to minimize learning effects. Two maximal effort trials will be performed with a 30-second rest between trials and the average of the trials (recorded in kg) will be used for data analysis. Additionally, subject body weight in kg will be recorded to allow for normalization of strength measures by dividing by subject body weight.
Change in lower trapezius force production | baseline and 1 minute after intervention
  A handheld dynamometer (HHD) (Hoggan MicroFET2) will be used to assess force production in standard MMT position using a "make test" as previously described. The "make test" will require the examiner to instruct the subject to slowly push into the HHD and increase their force production to a maximal level over a 5-second period of time. Prior to maximal isometric testing, a sub-maximal (50%) effort trial will be performed to minimize learning effects. Two maximal effort trials will be performed with a 30-second rest between trials and the average of the trials (recorded in kg) will be used for data analysis. Additionally, subject body weight in kg will be recorded to allow for normalization of strength measures by dividing by subject body weight.
Change in serratus anterior force production | baseline and 1 minute after intervention
  A handheld dynamometer (HHD) (Hoggan MicroFET2) will be used to assess force production in standard MMT position using a "make test" as previously described. The "make test" will require the examiner to instruct the subject to slowly push into the HHD and increase their force production to a maximal level over a 5-second period of time. Prior to maximal isometric testing, a sub-maximal (50%) effort trial will be performed to minimize learning effects. Two maximal effort trials will be performed with a 30-second rest between trials and the average of the trials (recorded in kg) will be used for data analysis. Additionally, subject body weight in kg will be recorded to allow for normalization of strength measures by dividing by subject body weight.

CONTACTS AND LOCATIONS:
Overall Officials: Jason K Grimes, PhD, Principal Investigator — Sacred Heart University

IPD SHARING:
Plan to Share IPD: Undecided
data regarding scapular kinematics during upper extremity elevation, pectoralis minor muscle length in standing, and force production in MMT positions for middle trapezius, lower trapezius, and serratus anterior; request for data should be made by email to: grimesj@sacredheart.edu

REFERENCES:
- [Background] Haik MN, Alburquerque-Sendin F, Silva CZ, Siqueira-Junior AL, Ribeiro IL, Camargo PR. Scapular kinematics pre- and post-thoracic thrust manipulation in individuals with and without shoulder impingement symptoms: a randomized controlled study. J Orthop Sports Phys Ther. 2014 Jul;44(7):475-87. doi: 10.2519/jospt.2014.4760. Epub 2014 May 22. PMID 24853923
- [Background] Muth S, Barbe MF, Lauer R, McClure PW. The effects of thoracic spine manipulation in subjects with signs of rotator cuff tendinopathy. J Orthop Sports Phys Ther. 2012 Dec;42(12):1005-16. doi: 10.2519/jospt.2012.4142. Epub 2012 Aug 17. PMID 22951537
- [Background] Kardouni JR, Pidcoe PE, Shaffer SW, Finucane SD, Cheatham SA, Sousa CO, Michener LA. Thoracic Spine Manipulation in Individuals With Subacromial Impingement Syndrome Does Not Immediately Alter Thoracic Spine Kinematics, Thoracic Excursion, or Scapular Kinematics: A Randomized Controlled Trial. J Orthop Sports Phys Ther. 2015 Jul;45(7):527-38. doi: 10.2519/jospt.2015.5647. Epub 2015 May 21. PMID 25996365
- [Background] Boyles RE, Ritland BM, Miracle BM, Barclay DM, Faul MS, Moore JH, Koppenhaver SL, Wainner RS. The short-term effects of thoracic spine thrust manipulation on patients with shoulder impingement syndrome. Man Ther. 2009 Aug;14(4):375-80. doi: 10.1016/j.math.2008.05.005. Epub 2008 Aug 15. PMID 18703377
- [Background] Strunce JB, Walker MJ, Boyles RE, Young BA. The immediate effects of thoracic spine and rib manipulation on subjects with primary complaints of shoulder pain. J Man Manip Ther. 2009;17(4):230-6. doi: 10.1179/106698109791352102. PMID 20140154
- [Background] Mintken PE, Cleland JA, Carpenter KJ, Bieniek ML, Keirns M, Whitman JM. Some factors predict successful short-term outcomes in individuals with shoulder pain receiving cervicothoracic manipulation: a single-arm trial. Phys Ther. 2010 Jan;90(1):26-42. doi: 10.2522/ptj.20090095. Epub 2009 Dec 3. PMID 19959652
- [Background] Leggin BG, Michener LA, Shaffer MA, Brenneman SK, Iannotti JP, Williams GR Jr. The Penn shoulder score: reliability and validity. J Orthop Sports Phys Ther. 2006 Mar;36(3):138-51. doi: 10.2519/jospt.2006.36.3.138. PMID 16596890
- [Background] Johnson MP, McClure PW, Karduna AR. New method to assess scapular upward rotation in subjects with shoulder pathology. J Orthop Sports Phys Ther. 2001 Feb;31(2):81-9. doi: 10.2519/jospt.2001.31.2.81. PMID 11232742
- [Background] Scibek JS, Carcia CR. Validation of a new method for assessing scapular anterior-posterior tilt. Int J Sports Phys Ther. 2014 Oct;9(5):644-56. PMID 25328827
- [Background] Watson L, Balster SM, Finch C, Dalziel R. Measurement of scapula upward rotation: a reliable clinical procedure. Br J Sports Med. 2005 Sep;39(9):599-603. doi: 10.1136/bjsm.2004.013243. PMID 16118295
- [Background] Borstad JD. Measurement of pectoralis minor muscle length: validation and clinical application. J Orthop Sports Phys Ther. 2008 Apr;38(4):169-74. doi: 10.2519/jospt.2008.2723. Epub 2007 Nov 21. PMID 18434665
- [Background] Michener LA, Boardman ND, Pidcoe PE, Frith AM. Scapular muscle tests in subjects with shoulder pain and functional loss: reliability and construct validity. Phys Ther. 2005 Nov;85(11):1128-38. PMID 16253043
- [Background] Michener LA, Kardouni JR, Sousa CO, Ely JM. Validation of a sham comparator for thoracic spinal manipulation in patients with shoulder pain. Man Ther. 2015 Feb;20(1):171-5. doi: 10.1016/j.math.2014.08.008. Epub 2014 Sep 6. PMID 25261090